CLINICAL TRIAL: NCT00581087
Title: Double-blind, Randomised, Placebo-controlled Phase III Study of Dehydroepiandrosterone (DHEA) in Respiratory Pulmonary Hypertension in Adults
Brief Title: Study of Dehydroepiandrosterone (DHEA) in Respiratory Pulmonary Hypertension in Adults
Acronym: DHEA-HTAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dromer; AFSSAPS 040479
Record Dates: First submitted 2007-12-26; First posted 2007-12-27 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypertension, Pulmonary
Keywords: Hypertension, pulmonary; DHEA; six-minute walk test; pulmonary arterial pressure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DHEA
  Interventions: Drug: DHEA treatment
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHEA treatment — DHEA : 200 mg/day hard gelatine capsule
  Arms: 1
Drug: Placebo — Treatment : 200 mg/day hard gelatine capsule
  Arms: 2

SUMMARY:
DHEA prevents and reverses chronic hypoxic pulmonary hypertension in a chronic hypoxic-pulmonary hypertension model in the rat. However, no study has been performed in human. The purpose of this study is to determine if DHEA is effective in the treatment of respiratory pulmonary hypertension in adults with Chronic Obstructive Pulmonary Disease (COPD) on exercise capacity and haemodynamic variables. Patients will receive after randomization either 200 mg oral DHEA or placebo over a one-year period. Evaluation concerns clinical parameters, echocardiography and right catheterization after and before treatment. Primary end-point is the six-minute walk test. This is a prospective double blind, randomized, placebo controlled study which will be realized in four university hospitals in France : Bordeaux, Strasbourg, Toulouse and Limoges.

Eight patients with pulmonary hypertension (New York Heart Association functional class III or IV) associated with COPD were included in a pilot study between 2004 and 2005. Inclusion criteria were: COPD was defined by FEV1/FVC < 70% of reference values; resting mean pulmonary artery pressure (assessment by right pulmonary catheterization) ≥ 25mmHg with mean pulmonary capillary wedge pressure ≤ 15mmHg, PaO2 ≤ 60mmHg at rest or PaO2 ≥ 60mmHg associated with significant fall in O2 saturation with exercise; oxygen treatment initiated more than six months previously. Exclusion criteria were: clinical or respiratory instability during the three months before the inclusion in the study; corticosteroids therapy (> 0.5mg/kg/day of prednisolone or as equivalent); hepatic (prothrombin time < 50%) or renal (creatininemia > 130µmol/L) failure; diabetes; left ventricular dysfunction; PSA (prostatic antigens > 2,5ng/ml) and past history or diagnosis of cancer. The study was conducted in accordance with the Good Clinical Practices Guidelines. The study protocol was approved by the ethics review board of the University Hospital of Bordeaux (France). Written informed consent was obtained for all patients and investigations were conducted according to the institutional guidelines and to the Helsinki principles. This trial conducted enrollment between 2004 and 2005, but had not been registered in ClinicalTrials.gov because it preceded this policy.(Study design: The dose of oral DHEA administered was 200 mg once daily for three months. At baseline and after three months of treatment, clinical evaluation included 6MWT, Borg dyspnea index, systolic and diastolic blood pressure, right heart catheterisation, lung function testing and serum DHEA levels were performed.)

DETAILED DESCRIPTION:
• Principal Objective : Efficacy of DHEA on exercise capacity (six-minute walk test)

* Secondary Objective :

  * Efficacy of DHEA on pulmonary arterial pressures (mean, systolic and diastolic), on systemic arterial pressures, pulmonary vascular resistances
  * Safety of DHEA treatment
  * Observance of treatment by DHEA
* Study design :

Double-blind, randomized, placebo-controlled Phase III study. Patients will be randomized into two parallel groups to receive either 200 mg oral DHEA or placebo over a one-year treatment. This is a multicentric study in the departments of respiratory medicine of Bordeaux, Strasbourg, Limoges and Toulouse (France).

• Inclusion criteria :

* Age ≥ 18 years old and ≤ 75 years old (*)
* Chronic Obstructive Pulmonary Disease with VEMS/CV < 70% ( **)
* Respiratory pulmonary hypertension with mean pulmonary arterial pressure ≥ 25 mmHg (**) related to normal pulmonary capillary pressure assessed by catheterization of the right side of the heart (pulmonary capillary wedge pressure ≤12mmHg)
* PO2 ≤ 60 mmHg assessed by arterial gazometry at ease (**) or PO2 > 60 mmHg, but related with high hypoxemia after exercise (six-minute walk test )
* Oxygenotherapy more than 6 months before pre-screening
* Written informed consent

(*) Inclusion of young adults concerns COPD related to asthma or cystic fibrosis (**) Criteria assessed from last health check or the last exams for COPD diagnosis

* Exclusion criteria :

  * Clinical instability and/or respiratory exacerbation within the previous three months
  * Clinical instability and/or respiratory exacerbation dangerous for catheterization
  * Pregnancy (ßHCG > 20 UI /l) or breastfeeding on going
  * General corticotherapy > 0,5 mg/kg/j prédnisolone equivalent
  * Hepatic insufficiency (TP < 50%) or renal insufficiency (creatininemia > 130 µmol/l) or diabetes mellitus type I or II (treated by oral antidiabetic oral or insulin)
  * Left-heart failure (coronary heart disease and/or left valvulopathy)
  * High level of prostatic specific antigen (PSA) (> 2,5ng/ml)
  * Previous cancer or treatment on going
* Study plan:

After the screening evaluation and written consent document, patients will be randomized into two groups placebo or DHEA, over a one year treatment.

• Number of subjects : 60 patients based on the increase of 30 % of the primary end-point, (six-minute walk test), i.e., 30 patients will be included in each group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years old (*)
* Chronic Obstructive Pulmonary Disease with FEVs/VC < 70% (**)
* Respiratory pulmonary hypertension with mean pulmonary arterial pressure ≥ 25 mmHg (**) related to normal pulmonary capillary pressure assessed by catheterization of the right side of the heart (pulmonary capillary wedge pressure ≤12mmHg)
* PO2 ≤ 60 mmHg assessed by arterial gazometry at ease (**) or PO2 > 60 mmHg, but related with high hypoxemia after exercise (six-minute walk test )
* Oxygenotherapy more than 6 months before pre-screening
* Written informed consent

(*) Inclusion of young adults concerns COPD related to asthma or cystic fibrosis (**) Criteria assessed from last health check or the last exams for COPD diagnosis

Exclusion Criteria:

* clinical instability and/or respiratory exacerbation within the previous three months
* clinical instability and/or respiratory exacerbation dangerous for catheterization
* Pregnancy (ßHCG > 20 UI /l) or breastfeeding on going
* General corticotherapy > 0,5 mg/kg/day prédnisolone equivalent
* Hepatic insufficiency (TP < 50%) or renal insufficiency (creatininemia > 130 µmol/l) or diabetes mellitus type I or II (treated by oral antidiabetic or insulin)
* Left-heart failure (coronary heart disease and/or left valvulopathy)
* High level of prostatic specific antigen (PSA) (> 2,5ng/ml)
* Cancer antecedent or treatment on going

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
six-minute walk test | inclusion and one year of treatment

SECONDARY OUTCOMES:
Pulmonary and systemic arterial pressures (mean, systolic and diastolic) | Inclusion and one after year of treatment
Pulmonary vascular resistances | Inclusion and after one year of treatment
Safety | along one year of treatment
Compliance | Along one year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claire Dromer, Dr, Principal Investigator — University Hospital, Bordeaux; Nicholas Moore, Pr, Study Chair — Universty Hospital, Bordeaux; Eric Dumas De La Roque, Dr, Study Director — University Hospital, Bordeaux
Locations (5):
- France (5):
  - University Hospital, Bordeaux, Bordeaux
  - APHP hospital Antoine Béclère GHU sud, Clamart
  - University Hospital, Limoges, Limoges
  - University Hospital, Strasbourg, Strasbourg
  - University Hospital, Toulouse, Toulouse

REFERENCES:
- [Background] Bonnet S, Dumas-de-La-Roque E, Begueret H, Marthan R, Fayon M, Dos Santos P, Savineau JP, Baulieu EE. Dehydroepiandrosterone (DHEA) prevents and reverses chronic hypoxic pulmonary hypertension. Proc Natl Acad Sci U S A. 2003 Aug 5;100(16):9488-93. doi: 10.1073/pnas.1633724100. Epub 2003 Jul 23. PMID 12878719
- [Derived] Dumas de La Roque E, Savineau JP, Metivier AC, Billes MA, Kraemer JP, Doutreleau S, Jougon J, Marthan R, Moore N, Fayon M, Baulieu EE, Dromer C. Dehydroepiandrosterone (DHEA) improves pulmonary hypertension in chronic obstructive pulmonary disease (COPD): a pilot study. Ann Endocrinol (Paris). 2012 Feb;73(1):20-5. doi: 10.1016/j.ando.2011.12.005. Epub 2012 Jan 26. PMID 22280813